CLINICAL TRIAL: NCT04382196
Title: The Impact of the COVID-19 Pandemic on Mental Health and Quality of Life of Healthcare Workers in a University Hospital
Brief Title: Impact of COVID-19 on Mental Health of Health Care Workers
Acronym: COVID-Impact
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-07564
Record Dates: First submitted 2020-05-08; First posted 2020-05-11 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Mental Health; Quality of Life
Keywords: Health care workers; Covid-19; Mental health
MeSH Terms: conditions — Psychological Well-Being; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health care workers: Health care workers at university hospital
  Interventions: Other: Online survey

INTERVENTIONS:
Other: Online survey — An online survey will be administered

SUMMARY:
The impact of the current Covid-19 pandemic on healthcare workers is enormous. This longitudinal study investigates the prevalence of mental health problems and the quality of life of healthcare workers during and after the Covid-19 pandemic. Underlying risk factors are also examined. Health care workers of the different Covid-19 cohort and transit wards, as well as the intensive care unit and (psychiatric) emergency services of the Ghent university hospital will be included, as well as the health care workers of 6 non-Covid-19 wards.

DETAILED DESCRIPTION:
The impact of the current Covid-19 pandemic on healthcare workers is enormous. Previous studies during the SARS outbreak demonstrated a significant burden and increase of mental health problems in health care workers.This longitudinal study aims to investigate the prevalence of mental health problems and the quality of life of health care workers during and after the Covid-19 pandemic. Health care workers of the different Covid-19 cohort and transit wards, as well as the intensive care unit and (psychiatric) emergency services of the Ghent university hospital will be included, as well as the health care workers of 6 non-Covid-19 wards. Participants will receive a monthly online survey during the government issued restrictions. After cessation of the restrictions participants will receive three-monthly surveys for a one-year-period.

Sociodemographic data, data regarding employment and previous mental health problems will be collected at the first survey. The Covid-19 status of the health care workers will be inquired at every survey. The Depression, Anxiety and Stress Scale (DASS-21), the Dutch translation of the Covid-19 Peritraumatic Distress Index (CPDI), the WHO Quality of Life-BREF (WHOQOL-BREF), and the Primary Care PTSD Screen for DSM-5 (PC-PTSD-5) and three items measuring social support will be administered at every survey.

ELIGIBILITY:
Inclusion Criteria:

* health care worker
* employed at inclusion at Covid cohort/transit or (psychiatric) emergency services or intensive care unit or 6 specified wards of the Ghent University Hospital

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All personnel of the above specified services of the university hospital involved in direct or indirect care will be eligible for inclusion
Sampling Method: Non-Probability Sample
Enrollment: 524 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms at baseline | Baseline
  Depressive symptoms as measured by the 7-item depression subscale of the self-reported 21-item Depression, Anxiety, and Stress Scale (DASS-21) (DASS-21-Depression). A higher score indicates more depressive symptoms with a minimum score of 0 and a maximum score of 21.
Change in depressive symptoms | Baseline, baseline + 30 days, baseline + 90 days, baseline + 180 days, baseline + 270 days, baseline + 360 days, baseline + 540 days, baseline + 900 days
  Depressive symptoms as measured by the 7-item depression subscale of the self-reported 21-item Depression, Anxiety, and Stress Scale (DASS-21) (DASS-21-Depression). A higher score indicates more depressive symptoms with a minimum score of 0 and a maximum score of 21.
Anxiety levels at baseline | Baseline
  Anxiety as measured by the 7-item anxiety subscale of the self-reported DASS-21 (DASS-21-Anxiety). A higher score indicates higher anxiety levels with a minimum score of 0 and a maximum score of 21.
Change in anxiety levels | Baseline, baseline + 30 days, baseline + 90 days, baseline + 180 days, baseline + 270 days, baseline + 360 days, baseline + 540 days, baseline + 900 days
  Anxiety as measured by the 7-item anxiety subscale of the self-reported DASS-21 (DASS-21-Anxiety). A higher score indicates higher anxiety levels with a minimum score of 0 and a maximum score of 21.
Stress levels at baseline | Baseline
  Stress as measured by the 7-item stress subscale of the self-reported DASS-21 (DASS-21-Stress). A higher score indicates higher stress levels with a minimum score of 0 and a maximum score of 21.
Change in stress levels | Baseline, baseline + 30 days, baseline + 90 days, baseline + 180 days, baseline + 270 days, baseline + 360 days, baseline + 540 days, baseline + 900 days
  Stress as measured by the 7-item stress subscale of the self-reported DASS-21 (DASS-21-Stress). A higher score indicates higher stress levels with a minimum score of 0 and a maximum score of 21.
Quality of life at baseline | Baseline
  Quality of life will be measured by the WHO Quality of Life Bref Questionnaire (WHOQOL-BREF). This self-report questionnaire has a minimum score of 0 and a maximum score of 100 with a higher score indicating higher quality of life. It includes different domains such as physical health, psychological health, social relationships and environment as well as two specific questions regarding an individual's overall perception of quality of life and physical health.
Change in Quality of life | Baseline, baseline + 30 days, baseline + 90 days, baseline + 180 days, baseline + 270 days, baseline + 360 days, baseline + 540 days, baseline + 900 days
  Quality of life will be measured by the WHO Quality of Life Bref Questionnaire (WHOQOL-BREF). This self-report questionnaire has a minimum score of 0 and a maximum score of 100 with a higher score indicating higher quality of life. It includes different domains such as physical health, psychological health, social relationships and environment as well as two specific questions regarding an individual's overall perception of quality of life and physical health.
Covid-19 related psychological distress | baseline
  Specific distress regarding Covd-19 will be measured by the Dutch translation of the COVID-19 Peritraumatic Distress Index (CPDI). This self-reported questionnaire inquires about the frequency of anxiety, depression, specific phobias, cognitive change, avoidance and compulsive behaviour, physical symptoms and loss of social functioning in the past week. The score ranges from 0 to 100, with higher scores indicating more distress.
Change in Covid-19 related psychological distress | Baseline, baseline + 30 days, baseline + 90 days, baseline + 180 days, baseline + 270 days, baseline + 360 days, baseline + 540 days, baseline + 900 days
  Specific distress regarding Covd-19 will be measured by the Dutch translation of the COVID-19 Peritraumatic Distress Index (CPDI). This self-reported questionnaire inquires about the frequency of anxiety, depression, specific phobias, cognitive change, avoidance and compulsive behaviour, physical symptoms and loss of social functioning in the past week. The score ranges from 0 to 100, with higher scores indicating more distress.
Post traumatic stress symptoms | Baseline
  The Primary Care PTSD Screen for DSM-5 (PC-PTSD-5) is a 5-item screen that was designed for use in primary care settings. The measure begins with an item designed to assess whether the respondent has had any exposure to traumatic events. If a respondent denies exposure, the PC-PTSD-5 is complete with a score of 0. However, if a respondent indicates that they have experienced a traumatic event over the course of their life, the respondent is instructed to respond to five additional yes/no questions about how that trauma exposure has affected them over the past month. The minimum score is 0 and the maximum score is 5 with higher scores indicating more PTSD-related symptoms.
Change in post traumatic stress symptoms | Baseline, baseline + 30 days, baseline + 90 days, baseline + 180 days, baseline + 270 days, baseline + 360 days, baseline + 540 days, baseline + 900 days
  The Primary Care PTSD Screen for DSM-5 (PC-PTSD-5) is a 5-item screen that was designed for use in primary care settings. The measure begins with an item designed to assess whether the respondent has had any exposure to traumatic events. If a respondent denies exposure, the PC-PTSD-5 is complete with a score of 0. However, if a respondent indicates that they have experienced a traumatic event over the course of their life, the respondent is instructed to respond to five additional yes/no questions about how that trauma exposure has affected them over the past month. The minimum score is 0 and the maximum score is 5 with higher scores indicating more PTSD-related symptoms.

SECONDARY OUTCOMES:
Perceived social support at baseline | Baseline
  Social support (from colleagues and employer) as perceived by participants will be measured by three items as measured on a 5-point Likert scale. For each item the minimum score is 1 and the maximum score is 5.
Change in perceived social support | Baseline, baseline + 30 days, baseline + 90 days, baseline + 180 days, baseline + 270 days, baseline + 360 days, baseline + 540 days, baseline + 900 days
  Social support (from colleagues and employer) as perceived by participants will be measured by three items as measured on a 5-point Likert scale. For each item the minimum score is 1 and the maximum score is 5.

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Lemmens, Study Director — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided